CLINICAL TRIAL: NCT04191980
Title: Multi-zone Computer-aided Prostate Segmentation on MR Images Using a Deep Learning-based Approach
Brief Title: Deep Learning for Prostate Segmentation
Acronym: GOPI-Segm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: GOPI-Segmentation_2019
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Prostate Cancer
Keywords: prostate segmentation; MR images
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Patients with a MRI on a 3 Tesla (T) unit: The total validation cohort is composed of axial T2-weighted images of the prostate obtained from 31 prostate MRIs on a 3T unit randomly chosen among the prostate MRIs performed at the Hospices Civils de Lyon in 20162015-2019
  Interventions: Other: Comparison of prostate multi-zone segmentation obtained with an automatic deep learning-based algorithm and two expert radiologists
- Patients with a MRI on a 1.5 Tesla unit: The total validation cohort is composed of axial T2-weighted images of the prostate obtained from 31 prostate MRIs on a 1.5T unit randomly chosen among the prostate MRIs performed at the Hospices Civils de Lyon in 20162015-2019
  Interventions: Other: Comparison of prostate multi-zone segmentation obtained with an automatic deep learning-based algorithm and two expert radiologists

INTERVENTIONS:
Other: Comparison of prostate multi-zone segmentation obtained with an automatic deep learning-based algorithm and two expert radiologists — The algorithm is used to perform a multizone segmentation of the prostate including delineation of : the whole prostate contours, the transition zone contours, the anterior fibromuscular stroma.
  The contours is independently corrected by 2 radiologists. The corrected contours of the different zones will be stored and for each zone 6 different metrics will be used to evaluate the difference between the initial and corrected contours:
  * Mean Mesh Distance: Average Boundary Distance (ABD) for each point of the reference segmentation. The distance to the closest point of the compared segmentation is first computed. Then the average of all these distances is computed and gives the ABD
  * General Hausdorff distance (HD)
  * 95% percentile (P) of the HD and the 95th (P) of the asymmetric HD distribution
  * 95% HD modified (HD95_1): different approach by first computing the 95th (P) of the asymmetric HD then taking the maximum
  * Dice coefficient
  * Difference in volumes

SUMMARY:
Because the diagnostic criteria for prostate cancer are different in the peripheral and the transition zone, prostate segmentation is needed for any computer-aided diagnosis system aimed at characterizing prostate lesions on magnetic resonance (MR) images. Manual segmentation is time consuming and may differ between radiologists with different expertise. We developed and trained a convolutional neural network algorithm for segmenting the whole prostate, the transition zone and the anterior fibromuscular stroma on T2-weighted images of 787 MRIs from an existing prospective radiological pathological correlation database containing prostate MRI of patients treated by prostatectomy between 2008 and 2014 (CLARA-P database).

The purpose of this study is to validate this algorithm on an independent cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* Prostate MRI contained in the PACS of the Hospices Civils de Lyon
* Performed in 2016-2019

Exclusion Criteria:

* MRIs from patients who already had treatment for prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Random selection in the Picture Archiving and Communication System (PACS) of the Hospices Civils de Lyon among examinations performed between 2016 and 2019
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Mean Mesh Distance (Mean) between the contours of the whole prostate made by the algorithm and the two radiologists | Month 11
  The Mean Mesh Distance corresponds to the Average Boundary Distance (ABD) for each point of the reference segmentation. The distance to the closest point of the compared segmentation is first computed. Then the average of all these distances is computed and gives the ABD.
  The Mean Mesh Distance between the contours of the whole prostate made by the algorithm and each radiologist will be used as primary outcome measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot, Lyon, France